CLINICAL TRIAL: NCT04633265
Title: ECG-I Targeted Ablation for Persistent AF Not Responding to Pulmonary Vein Isolation: Results of a Two Staged Strategy (ECG-I TARGET AF2)
Brief Title: ECG-I Targeted Ablation for Persistent AF Not Responding to Pulmonary Vein Isolation Results of a Two Staged Strategy.
Acronym: TARGET-AF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218367-3
Record Dates: First submitted 2018-07-10; First posted 2020-11-18 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation ECG-I Mapping Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ECG-I Mapping and Ablation of drivers (Experimental): ECG-I Mapping will be performed and drivers will be ablated as directed by ECG-I.
  Interventions: Device: ECG-I Mapping of Atrial Fibrillation

INTERVENTIONS:
Device: ECG-I Mapping of Atrial Fibrillation — Catheter ablation of Atrial Fibrillation guided by ECG-I

SUMMARY:
Atrial Fibrillation (AF) is a irregular heart rhythm associated with significant morbidity and mortality. Catheter ablation is a treatment where catheters are passed through the veins in the leg into the left atrium of the heart and lines of scar is delivered to disrupt tissue causing and maintaining atrial fibrillation. Current strategies involve isolating the pulmonary veins which have been shown to trigger and maintain AF. However, success rates for persistent AF lie in the region of 30-60% due to the drivers of AF residing elsewhere to the Pulmonary Veins antra.

The ECG-I is a system which involves wearing a jacket with many ECG electrodes to record electrical activity from the surface of the body. A CT scan then shows where these electrodes are relative to the atria, and computer modelling is used to reconstruct the movements of electricity on the surface of the heart and therefore identifying where the drivers (tissue causing and maintaining AF) are located.

Unfortunately, not all patients respond to PVI due to the drivers of AF being located in areas other than within the Pulmonary Veins. Identifying the drivers of AF is very difficult and the role they play has yet to be proved scientifically.

PHENOTYPE AF is an ongoing clinical trial in which 100 patients with persistent AF are receiving cryoballoon pulmonary vein isolation for persistent AF (NCT03394404). Patients with recurrent AF or atrial tachycardia within 1 year following pulmonary vein isolation for AF within this trial will be recruited into this study. Up to 50 such patients who have failed Pulmonary Vein Isolation will be enrolled. These patients will undergo a second procedure at which time participants will undergo catheter ablation of drivers of AF and will then be followed up for 12 months.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is the commonest heart rhythm disturbance and is associated with significant morbidity and mortality. Catheter ablation (CA) is a procedure where catheters (leads) are passed into the heart and energy is used to disrupt and isolate (by freezing or cauterising) heart tissue causing AF. CA is an established therapy for AF. Success rates for CA for paroxysmal AF lies in the region of 70% or better. However, success rates for persistent AF is much lower and estimates lie in the region of 30-60%.

Current CA protocols for AF centre on isolating the pulmonary veins (the pulmonary veins drain into the left atrium) which have been proven to trigger AF. Pulmonary Vein Isolation (PVI) ablation alone seems sufficient to remove the trigger for the vast majority of patients with paroxysmal AF. However, in patients with persistent AF it is common for AF to continue after the pulmonary veins have been electrically isolated.

The difference in success rates between the paroxysmal and persistent form of AF is thought to be due to changes within the heart atria after AF has been established for some time. In persistent AF the atria dilate and remodel structurally and electrically, and therefore the maintenance of persistent AF differs from paroxysmal AF.

Persistent AF is thought to be maintained by focal sources, whether rotors or sites of radial activation. Currently, targeting other sites within the atria in addition to PVI such as fractionated electrograms (areas of electrical activity) are thought to be imprecise and require extensive ablation. Often AF will persist despite targeting additional sites within the atria.

One particular challenge is to select patients likely to benefit from CA. CA carries an approximate less than 1% risk of life threatening complication. Therefore being able to select suitable patients is desirable in order to prevent unnecessary procedures.

Currently clinical characteristics of patients or structural imaging have limited accuracy in selecting patients likely to benefit from CA. Mapping studies have shown that patients with persistent AF who have higher frequency signals near the pulmonary veins than being distributed in the left atrial body are more likely to terminate to sinus rhythm (normal heart rhythm) with PVI alone and to maintain sinus rhythm.

Studies have suggested that patients undergoing standard PVI ablation procedures for persistent AF who have coincidental interruption of drivers have a far better long term outcome. This suggests that the characteristics of atrial heart tissue and electrical activation patterns maintaining AF are likely to determine the response to ablation therefore it may be possible to determine more directly and accurately the likelihood of success by performing non-invasive mapping of the atria using the ECG-I.

ECG-I is able to localise the drivers of AF and one of the objectives is to study the electrical characteristics of the tissue. ECG-I is currently being used in research into AF. A recently published a study using ECG-I to identify targets of ablation in 103 patients. The on-going multicentre AFACART study has published early data to suggest that ECG-I can identify the drivers of AF and improve CA success rates.

PHENOTYPE AF is an ongoing clinical trial in which 100 patients with persistent AF are receiving cryoballoon pulmonary vein isolation for persistent AF (NCT03394404). Patients with recurrent AF or atrial tachycardia within 1 year following pulmonary vein isolation for AF within this trial will be recruited into this study. Up to 50 such patients who have failed Pulmonary Vein Isolation will be enrolled. These patients will undergo a second procedure at which time participants will undergo catheter ablation of drivers of AF and will then be followed up for 12 months.

ELIGIBILITY:
Patients with recurrent AF or atrial tachycardia within 1 year of ablation for persistent AF in the PHENOTYPE AF trial (NCT03394404). Original inclusion criteria for PHENOTYPE AF trial:

* Persistent AF (i.e. episodes of AF that are continuous for > 1 week)
* Willing for ablation.
* Age between 18 to 80.

Exclusion Criteria:

* Exclusions:

  * Continuous persistent AF > 2 years duration
  * Left atrial diameter > 5 cm
  * Severe left ventricular impairment (EF < 40%)
  * New York Heart Association class 3 or 4 heart failure
  * Known hypertrophic cardiomyopathy, cardiac sarcoid or Arrhythmogenic Cardiomyopathy.
  * Known inherited arrhythmia such as Brugada or long QT syndromes
  * Valvular disease that is more than moderate
  * History of valve replacement (metallic or tissue)
  * History of congenital heart disease (other than patent foramen ovale)
  * Previous left atrial ablation (percutaneous or surgical)
  * Cardiac surgery or percutaneous coronary intervention within the last 3 months.
  * Myocardial infarction or unstable angina within the last 3 months.
  * Unwillingness for ablation
  * Unwillingness to be involved in study
  * Suspected reversible cause of AF
  * Any other contraindication to catheter ablation
  * Age < 18 yrs or > 80 years
  * Pregnancy
  * Morbid obesity (defined as body mass index >40)
  * Any other medical problem likely to cause death within the next 18 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants free from Atrial Arrhythmia at 12 months | 12 months
  Number of participants free from atrial arrhythmia (including both AF and atrial tachycardia) at 12 months following their procedure

SECONDARY OUTCOMES:
Rates of termination of AF with ECGI guided ablation | Intra-procedural (day 1)
  The proportion of patients in whom AF terminates with ablation during the catheter ablation procedure
Number of participants free from AF at 12 months | 12 months
  Number of participants free from AF at 12 months following their procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided